CLINICAL TRIAL: NCT03713047
Title: A National Center for Persistent Severe Pain After Groin Hernia Repair: Five-year Prospective Data
Brief Title: A National Center for Persistent Severe Pain After Groin Hernia Repair
Acronym: Q5Y
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, mads u werner, Principal Investigator, University of Copenhagen
Other Study IDs: H-2-2011-023
Record Dates: First submitted 2018-07-19; First posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Inguinal Hernia; Chronic Pain
Keywords: Questionnaire; Long term follow up; Surgical Procedure; Groin hernia repair; Neuropathy; Inflammation; Chronic pain; ADL-functions; Psychometrics; Quantitative sensory testing (QST)
MeSH Terms: conditions — Hernia, Inguinal; Chronic Pain; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, consecutive cohort study presents nationwide 5-year outcome data on patients with severe persistent pain after groin hernia repair (SPG).

The inclusion criteria were SPG-related impairment of physical and social life. Two-hundred-four out of 222 patients (92%) were analyzed. Relevant surgical records were obtained, and examinations were by standardized clinical and neurophysiological tests. Patients demonstrating pain sensitivity to pressure algometry in the groin were evaluated regarding exploratory surgery, while patients with putative neuropathic pain received pharmacotherapy. Questionnaires at baseline (Q0) and five-year (Q5Y) were used in outcome-analyses of pain-intensity (numeric rating scale [NRS] 0-10) and the pain-related effect on the activity-of-daily-living (Activities Assessment Scale, AAS).

DETAILED DESCRIPTION:
Severe persistent pain after groin hernia repair (SPG) causes psychophysical disability and impairs quality-of-life for a considerable number of individuals each year.1-3 In the United States, 600,000 groin hernia repairs (GHR) are performed annually, and a conservative estimate is that 2%, corresponding to 12,000 individuals, each year will develop this debilitating pain condition.4 The management of SPG remains a daunting challenge to the medical profession 5, often requiring multidisciplinary efforts.1,6 Several surgical procedures have indicated substantial pain-relieving effects in SPG1,7 however few well-powered, controlled studies have been presented.8,9 In pharmacological and neuromodulation procedures, most studies are still case-based or uncontrolled.

In 2010, the authors established a dedicated tertiary center for SPG-patients open for referral on a nationwide basis. The objectives were, first, to analyze the pathophysiological mechanism behind the pain, second, to implement optimal medical and surgical pain management and third, to perform clinical SPG-research projects. Standardized clinical and neurophysiological tests guided the management paradigm for each patient. Treatment outcomes were evaluated prospectively using baseline questionnaires (Q0) and a 5-year questionnaire (Q5Y) mailed at the end of 2014 to all patients referred to the center.

The focus of the present study is first, to present clinical, neurophysiological and psychometric data on SPG-patients at referral, and second, to evaluate and compare efficacies of exploratory surgical and non-surgical treatment, based on a consecutive follow-up cohort of 222 patients.

ELIGIBILITY:
Inclusion Criteria:

* Severe persistent pain after groin hernia repair (activity-related or maximal pain intensity > 7 NRS-units [numeric rating scale 0-10])
* Severe persistent pain after groin hernia repair-related serious impairment of working and social life.

Exclusion Criteria:

* Minors or persons of legally incompetence
* Participants, who do not speak or understand Danish
* Participants, who cannot cooperate with the investigator or the examination procedure
* Recurrent hernia
* Known neurological disease or disorders in the groin area of other origin
* Psychiatric disease
* Abuse of alcohol or drugs - according to investigator's evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe persistent pain after groin hernia repair with psychophysical disability referred to the dedicated tertiary center for these patients on a nationwide basis.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 2010-2015
  Numeric Rating Scale (NRS; 0-10 units)
Activity of Daily Living (ADL) score | 2010-2015
  Activities Assessment Scale (AAS; 8 specified physical activities; 0-8 units each)

SECONDARY OUTCOMES:
Assessments of Anxiety and Depression | 2010-2015
  Hospital Anxiety and Depression Scale (HADS; 14 item scale; 0-21 units)
Assessment of Pain Catastrophizing | 2010-2015
  Pain Catastrophizing Scale (PCS; 13 item scale; 0-65 units)

CONTACTS AND LOCATIONS:
Overall Officials: Mads U Werner, MD, PhD, Principal Investigator — Neuroscience Center, Copenhagen University Hospital, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available as a supplement to the published scientific article.

REFERENCES:
- [Background] Werner MU. Management of persistent postsurgical inguinal pain. Langenbecks Arch Surg. 2014 Jun;399(5):559-69. doi: 10.1007/s00423-014-1211-9. Epub 2014 May 23. PMID 24849039
- [Background] Nikkolo C, Kirsimagi U, Vaasna T, Murruste M, Suumann J, Seepter H, Lepner U. Prospective study evaluating the impact of severity of chronic pain on quality of life after inguinal hernioplasty. Hernia. 2017 Apr;21(2):199-205. doi: 10.1007/s10029-016-1569-4. Epub 2016 Dec 26. PMID 28025741
- [Background] Niccolai P, Ouchchane L, Libier M, Beouche F, Belon M, Vedrinne JM, El Drayi B, Vallet L, Ruiz F, Biermann C, Duchene P, Chirat C, Soule-Sonneville S, Duale C, Dubray C, Schoeffler P. Persistent neuropathic pain after inguinal herniorrhaphy depending on the procedure (open mesh v. laparoscopy): a propensity-matched analysis. Can J Surg. 2015 Apr;58(2):114-20. doi: 10.1503/cjs.008314. PMID 25799247
- [Background] Cohen SP, Raja SN. Prevention of chronic postsurgical pain: the ongoing search for the holy grail of anesthesiology. Anesthesiology. 2013 Feb;118(2):241-3. doi: 10.1097/ALN.0b013e31827d4129. No abstract available. PMID 23340346
- [Background] Kehlet H, Roumen RM, Reinpold W, Miserez M. Invited commentary: Persistent pain after inguinal hernia repair: what do we know and what do we need to know? Hernia. 2013 Jun;17(3):293-7. doi: 10.1007/s10029-013-1109-4. Epub 2013 May 21. No abstract available. PMID 23686405
- [Background] Chen DC, Hiatt JR, Amid PK. Operative management of refractory neuropathic inguinodynia by a laparoscopic retroperitoneal approach. JAMA Surg. 2013 Oct;148(10):962-7. doi: 10.1001/jamasurg.2013.3189. PMID 23903521
- [Background] Magnusson N, Gunnarsson U, Nordin P, Smedberg S, Hedberg M, Sandblom G. Reoperation for persistent pain after groin hernia surgery: a population-based study. Hernia. 2015 Feb;19(1):45-51. doi: 10.1007/s10029-014-1340-7. Epub 2014 Dec 18. PMID 25519077
- [Background] Nikkolo C, Lepner U. Chronic pain after open inguinal hernia repair. Postgrad Med. 2016 Jan;128(1):69-75. doi: 10.1080/00325481.2016.1121090. Epub 2015 Dec 4. PMID 26567717
- [Background] Kehlet H, Bay-Nielsen M; Danish Hernia Database Collaboration. Nationwide quality improvement of groin hernia repair from the Danish Hernia Database of 87,840 patients from 1998 to 2005. Hernia. 2008 Feb;12(1):1-7. doi: 10.1007/s10029-007-0285-5. Epub 2007 Oct 16. PMID 17939015
- [Background] McCarthy M Jr, Jonasson O, Chang CH, Pickard AS, Giobbie-Hurder A, Gibbs J, Edelman P, Fitzgibbons R, Neumayer L. Assessment of patient functional status after surgery. J Am Coll Surg. 2005 Aug;201(2):171-8. doi: 10.1016/j.jamcollsurg.2005.03.035. PMID 16038812
- [Background] Aasvang EK, Gmaehle E, Hansen JB, Gmaehle B, Forman JL, Schwarz J, Bittner R, Kehlet H. Predictive risk factors for persistent postherniotomy pain. Anesthesiology. 2010 Apr;112(4):957-69. doi: 10.1097/ALN.0b013e3181d31ff8. PMID 20234307
- [Background] Bischoff JM, Koscielniak-Nielsen ZJ, Kehlet H, Werner MU. Ultrasound-guided ilioinguinal/iliohypogastric nerve blocks for persistent inguinal postherniorrhaphy pain: a randomized, double-blind, placebo-controlled, crossover trial. Anesth Analg. 2012 Jun;114(6):1323-9. doi: 10.1213/ANE.0b013e31824d6168. Epub 2012 Mar 30. PMID 22467891
- [Background] Aasvang EK, Kehlet H. Persistent sensory dysfunction in pain-free herniotomy. Acta Anaesthesiol Scand. 2010 Mar;54(3):291-8. doi: 10.1111/j.1399-6576.2009.02137.x. Epub 2009 Oct 15. PMID 19839945
- [Derived] Jensen EK, Ringsted TK, Bischoff JM, Petersen MA, Rosenberg J, Kehlet H, Werner MU. A national center for persistent severe pain after groin hernia repair: Five-year prospective data. Medicine (Baltimore). 2019 Aug;98(33):e16600. doi: 10.1097/MD.0000000000016600. PMID 31415351